CLINICAL TRIAL: NCT00740987
Title: Evaluation of Intermittent Pneumatic Compression Associated With Elastic Stockings and Anticoagulant Prophylaxis Versus Anticoagulant Prophylaxis Alone on Venous Thromboembolism Incidence in ICU Patients Without High Risk of Bleeding
Brief Title: Efficacy of the Association Mechanical Prophylaxis + Anticoagulant Prophylaxis on Venous Thromboembolism Incidence in Intensive Care Unit (ICU)
Acronym: CIREA2
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University Hospital, Brest (Other)
Collaborators: Tyco Healthcare Group (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CIREA2
Record Dates: First submitted 2008-08-22; First posted 2008-08-25 (Estimated); Last update posted 2015-02-11 (Estimated); Status verified 2014-12

CONDITIONS: No High Risk of Hemorrhage
Keywords: Mechanical device; Intermittent pneumatic compression; Venous thromboembolism prophylaxis; Intensive care unit; Hospitalization; Intensive; Care; Unit

ARMS (2):
- 1 (No Intervention): No Intermittent pneumatic compression of the lower limbs during hospitalisation in reanimation unit
- 2 (Experimental): Intermittent pneumatic compression of the lower limbs during hospitalisation in reanimation unit
  Interventions: Device: Intermittent pneumatic compression of the lower limbs

INTERVENTIONS:
Device: Intermittent pneumatic compression of the lower limbs — No Intermittent pneumatic compression of the lower limbs during hospitalisation in reanimation unit
  Arms: 2

SUMMARY:
This multicentre open-label randomized parallel-group trial aims to compare the association of intermittent pneumatic compression of the lower limbs + elastic stockings + anticoagulant prophylaxis to anticoagulant prophylaxis alone on the incidence of venous thromboembolism systematically evaluated at day 6, in patients hospitalized in intensive care units and without high bleeding risk.

DETAILED DESCRIPTION:
Background: Venous thromboembolism is a leading cause of morbi-mortality for patients hospitalized in intensive medical care units. Nevertheless, few studies evaluating prophylactic methods exist. Data from these studies demonstrate however that unfractionated heparin and low molecular weight heparin are effective to reduce the incident rate of asymptomatic deep venous thrombosis (DVT) of the lower limbs by 50 % compared to the absence of prophylaxis. Rate of asymptomatic DVT remains about 15 %. Mechanical devices such as elastic stockings (ES) or intermittent pneumatic compression (IPC), devoid of bleeding risk, can be associated with heparins, with good efficacy in some specific clinical settings. The effect of combined treatment use has never been evaluated rigorously in intensive medical care units.

Objective:

To compare the association IPC+ ES + anticoagulant prophylaxis to anticoagulant prophylaxis alone in patients without high bleeding risk and hospitalized in medical intensive care units on symptomatic or asymptomatic venous thromboembolism incidence, evaluated systematically at day 6.

Design: Multicentre open-label randomized parallel-group trial with blinded evaluation of outcomes, and an inclusion period of 24 month. Brest CIC (Centre d'Investigations cliniques, research center) coordinates this multicentre trial.

Outcomes:

The primary endpoint is a combined criterion (blindly evaluated) between day 1 and day 6:

1) Non fatal symptomatic venous thromboembolic event (objectively confirmed) between day 1 and day 6, 2) death due to a pulmonary embolism between day 1 and day 6, and 3) asymptomatic DVT detected by ultrasonography systematically done at day 6.

Patients number:

Assuming a DVT frequency of 10 % in the control group (anticoagulant prophylaxis alone), we calculated that 1436 patients will be required for the study to have 80% power to detect a 40 % reduction in the relative risk with a two-sided alpha level of 5%. Because of about 20 % deaths in the first days, we decide to increase the number at 1580 subjects.

Statistical analysis:

Efficacy analysis is performed on an 'intention-to-treat' basis. The frequencies of the combined primary outcome at day 6 are compared between groups using an exact one-sided Fischer test. Adjustment for stratification variables used Cochran-Mantel-Haenszel test. Relative risk and absolute risk reduction are computed with their 95% CIs. A logistic regression model is used to take into account potential imbalance in baseline characteristics.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 Years,
* Admission in intensive medical care unit
* No high risk for hemorrhage in CIREA 2
* Written informed consent given by the patient or relative.

High risk for hemorrhage is defined by:

* symptomatic bleeding or organic lesions likely to bleed,
* hemophilic diseases,
* haemostatic abnormalities: platelet count < 50 000/mm 3, APTT > 2 N, prothrombin time < 40%,
* recent intra-cerebral hemorrhage,
* severe anemia (Hemoglobin < 7 g/dl) due to a bleeding or unexplained.

Exclusion Criteria:

* Age < 18 years,
* Patient refusal,
* Admission in intensive care unit ≥ 36 hours
* Admission in intensive care unit likely for < 72 hours
* A "do not resuscitate" order
* IPC contra-indication: Recent DVT (< 3 month), severe lower limbs arteriopathy (III and IV), any arterial graft of the legs, a wound in the lower limb related either to a vascular disease (ulcer) or a trauma.
* High risk for hemorrhage
* Patient who needs a curative anticoagulant treatment (DVT, PE, PE suspicion, atrial fibrillation, myocardial infarction, acute coronary syndrome…).
* Patients with anticoagulant prophylaxis contra-indication

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 621 (Actual)
Dates: Start 2007-10; Primary Completion 2015-01 (Actual); Study Completion 2015-01 (Actual)

PRIMARY OUTCOMES:
combined criterion evaluated at day 6 ± 2 days after randomization: symptomatic venous thromboembolic event, non fatal, objectively confirmed, Death related to PE, Asymptomatic DVT of the lower limbs detected by CUS on day 6. | 6 +/- 2 days

SECONDARY OUTCOMES:
Symptomatic thromboembolic events occurred between day 6 and day 90, and total mortality evaluated at 1 month and 3 months. | 6 days to 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Karine LACUT, MD, Study Director — CHU Brest France, Univ Brest, EA 3878
Locations (15):
- France (14):
  - CHU d'Angers, Angers
  - CH d'Angoulême, Angoulême
  - HIA Clermont-Tonnerre, Brest
  - Medical Intensive Care Unit, Brest
  - CH de Corbeil Essonne, Corbeil Essonne
  - CHU de Dijon, Dijon
  - Medical Intensive Care Unit, Lille
  - CH Montauban, Montauban
  - CH de Morlaix, Morlaix
  - Medical Intensive Care Unit, Paris
  - CHU de Poitiers, Poitiers
  - CH de Quimper, Quimper
  - CH de St Malo, St-Malo
  - CHU de Tours, Tours
- CH Monaco, Monaco, Monaco